CLINICAL TRIAL: NCT04126460
Title: High-risk Recurrent or Second Primary HNSCC With PD-1 Antibody Adjuvant After Salvage Surgery: The RePASS Study
Brief Title: High-risk Recurrent or Second Primary HNSCC With PD-1 Antibody Adjuvant After Salvage Surgery(RePASS)
Acronym: RePASS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019HNRT02
Record Dates: First submitted 2019-10-12; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck; recurrent disease; PD-1; salvage surgery; Second Primary
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab (Experimental): Injection; dosage form: 6ml: 240mg; frequency: 240mgQ3W; duration: 17cycles (12 months) or randomization to the date of the first documented progression
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab is a type of PD-1 antibody
  Other Names: JS001

SUMMARY:
This is a non-randomized, phase II, open-label study. The goal of this clinical research study is to investigate the efficacy and safety of adjuvant Toripalimab in high-risk recurrent/secondary HNSCC after salvage surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically (histologically or cytologically) confirmed diagnosis of recurrent or second primary squamous cell carcinoma (SCC) of the head and neck. Known p16 status for oropharynx carcinoma.

  2.Patients must have had prior radiation for head and neck SCC with ≥ 75% of the present tumor volume in areas that have been previously irradiated to at least 45 Gy or the intersection between the first irradiation and the reirradiation fields had to be greater than 65%.

  3. Patients with at least one high risk factors after salvage surgery ①positive margin; ②close margin（<5mm); ③ENE;④PNI;⑤LVI; ⑤ rStaging III-IV( AJCC 8th).

  4. No macroscopic residual disease after salvage surgery.

  5.No distant metastasis.

  6.Eastern Cooperative Oncology Group Performance Status (ECOG) performance scale: 0-1.

  7.Adequate organ and bone marrow function: CBC: absolute neutrophil count (ANC) ≥ 1.5 × 10^9 / L; platelet count (PLT) ≥ 80 × 10^9 / L; hemoglobin content (HGB) ≥ 8.0 g / dL.

Liver function: serum total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN.

Renal function: serum creatinine (Cr) ≤ 1.5 × ULN.

8.Female subject of childbearing potential should have a negative urine or serum pregnancy test < 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

9.Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of study therapy through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses > 1 year.

10.Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of the study therapy.

11.Voluntarily signed written informed consent form, willing and able to comply with scheduled visits and other requirements of the study.

Exclusion Criteria:

* 1. Women who are pregnant or lactating.

  2.Subjects with active, known or suspected autoimmune disease such as interstitial pneumonia, uveitis, Crohn's disease, autoimmune thyroiditis. Subjects with cured childhood asthma, type I diabetes mellitus and hypothyroidism only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment.

  3.Subjects who are using systemic immunosuppressive agents and continue the dose within 2 weeks prior to the enrollment.

  4.Is currently participating in and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to randomization.

  5.There have been other malignant tumors in the past 5 years, except the cured skin basal cell carcinoma, cervical carcinoma in situ and superficial bladder cancer.

  6.Prior therapy with anti-PD-1,anti-PD-L1,anti-CTLA4 antibody.

  7.Uncontrolled concomitant disease, including but not limited to : Active or poorly controlled severe infection Human Immunodeficiency Virus (HIV) infection (HIV antibody positive) Known acute or chronic active hepatitis B (HBV DNA positive) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection Active tuberculosis Symptomatic congestive heart failure (New York Heart Association grade III-IV) or symptomatic, poorly controlled arrhythmia Uncontrolled hypertension (SBP ≥ 160mmHg or DBP ≥ 100mmHg) Prior arterial thromboembolism event, including myocardial infarction, unstable angina, stroke, and transient ischemic attack, within 6 months of enrollment.

  8.Upon the judgment by the investigator, subjects have other factors that possibly cause the halfway-termination of this study, such as other serious illnesses (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, with family or social factors, which may influence the safety of the subject, or the collection of trial data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
1 year disease-free survival | 1 year
  from date of enrollment until date of first documented disease progression or death from any cause, assessed up to 1 year

SECONDARY OUTCOMES:
1 year overall survival | 1 year
  from date of enrollment until date of death from any cause, assessed up to 1 year
1 year local-regional recurrence-free survival | 1 year
  from date of enrollment until date of first documented local-regional recurrence or death from any cause, assessed up to 1 year
1 year distant metastasis-free survival | 1 year
  from date of enrollment until date of first documented distant metastasis or death from any cause, assessed up to 1 year
Treatment-related adverse events (AEs) | from the date of enrollment to 90 days after last dose of study treatment
  The grade of AEs and the number of patients with AEs are assessed by the investigator based on CTCAE v4.0 from the date of enrollment to 90 days after last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shengjin Dou, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided